CLINICAL TRIAL: NCT04336514
Title: A Longitudinal Quantitative Assessment of the Effectiveness of Metatarsal Pads on Plantar Pressures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Michener Institute for Education at UHN (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-5921
Record Dates: First submitted 2020-02-24; First posted 2020-04-07 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Forefoot Callus; Podiatry; Foot Dermatoses; Keratosis
MeSH Terms: conditions — Foot Dermatoses; Keratosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental)
  Interventions: Device: Semi-compressed felt pad (SCF)

INTERVENTIONS:
Device: Semi-compressed felt pad (SCF) — Participants with forefoot callus will receive routine treatment of debridement of callus. Along with the debridement, a Plantar Metatarsal Pad (PMP) made of Semi-Compressed Felt (SCF) with appropriate cut outs will be placed in their shoes. The thickness of the SCF would be selected based on the patient weight, and appropriateness of the thickness would be confirmed by the Medilogic pressure measurement. A 50% pressure reduction is the desired outcome.

SUMMARY:
Musculoskeletal deformities of the foot and abnormal biomechanics can create areas of high pressure over bony prominences on the plantar aspect of the foot and often lead to the formation of calluses and corns. Calluses and corns are reported to be the most prevalent foot conditions affecting peoples' lifestyles due to pain and disability. Redistribution of plantar pressure away from areas of high pressure offloading using felt pads to treat corns and calluses is a common practice in chiropody. A more comprehensive understanding of how rapidly the felt pads compress and become less effective in offloading pressure is needed to design better treatment plans to manage calluses and corns and improve patients' quality of life. The objectives of this study are: 1) develop a guideline which informs, at what duration (number of weeks) the semi compressed felt (SCF) Plantar Metatarsal Pad (PMP) should be replaced to manage plantar forefoot callus; 2) Test the guideline by replacing the SCF padding at the determined time interval. The study will be conducted at the Michener Chiropody Clinic at the Michener Institute of Education at UHN. In order to address patient selection bias, the investigators will be recruiting the first 25-40 participants presenting with forefoot callus who meet the inclusion criteria and consent to participate in the study. An exploratory, descriptive and analytic repeated measures study design will be used to address our research questions. The descriptive approach will provide insight into the nature of change over time in the dependent variables, pain and pressure, and an analytic approach will enable further insight into the relationship between those variables. The quantitative metrics used are average plantar pressure at the callus site, as well as self-reported pain using a Visual-Analog Scale (VAS). Results from the first phase will inform the development of the guideline for pad replacement, which in turn will be tested in the next phase of the study.

ELIGIBILITY:
Inclusion Criteria:

The participants to be studied are from the general population with callus on the plantar aspect of the forefoot. The participants must have appropriate footwear with adequate space for pads and must be agreeable to wearing them majority of the study period for weight bearing activities. Participants must be willing to attend clinic every two weeks for 8 weeks

Exclusion Criteria:

Participants with an active or past history of foot ulcers, those with Charcot neuroarthropathy as well as those who were unable to walk unaided will be excluded from the study. All participants will undergo a neuropathic assessment, including the vibration using a 127Hz tuning fork, protective sensation using a 10 gram monofilament and proprioception to exclude patients with neuropathy. Participants will be excluded if they have any foot skin disorders such as infections, dermatitis and psoriasis. Furthermore, anyone with neuropathy or diabetes for over 5 years will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in Average Plantar Pressure 0-8 weeks | Change from baseline to 8 weeks
  The change in the average value of plantar pressure identified during the gait cycle from baseline to 8 weeks after the application of the semi-compressed felt pad.

SECONDARY OUTCOMES:
Perceived pain | 0 (pre and post insertion of SCF), 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Self-reported levels of pain will be recorded using the Visual Analogue Scale (0-100)
Physical Activity | 0 (pre and post insertion of SCF), 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  23 item questionnaire assessing the daily activity profiles of the participants.
Sociodemographic data- employment | 0 (pre and post insertion of SCF), 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Location of place of employment - at home or outside of home
Sociodemographic data - job description | 0 weeks
  Brief description of job demands
Daily physical activity- workday sitting time | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Time spent sitting on a typical work day in hours
Daily physical activity- weekend sitting time | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Time spent sitting on a typical weekend day in hours
Daily physical activity- work day standing time | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Time spent standing on a typical work day in hours
Daily physical activity- weekend standing time | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Time spent standing on a typical weekend day in hours
Daily physical activity- workday walking time | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Time spent walking or running or climbing on a typical work day in hours
Daily physical activity- weekend walking time | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Time spent walking or running or climbing on a typical weekend day in hours
Daily physical activity- workday time spent on feet | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Category of time spent on feet in hours on a typical work day in hours
Daily physical activity- weekend time spent on feet | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Category of time spent on feet in hours on a typical weekend day in hours
Daily physical activity- workday strain on feet | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Category of foot strain experienced on a typical work day
Daily physical activity- weekend strain on feet | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Category of foot strain experienced on a typical weekend day
Daily physical activity- time of wearing pad on a workday | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Category of time for which pad was worn on a typical work day in hours
Daily physical activity- time of wearing pad on a weekend day | 0 weeks, 2 weeks, 4 weeks, 6 weeks, and 8 weeks
  Category of time for which pad was worn on a typical weekend day in hours

CONTACTS AND LOCATIONS:
Overall Officials: Ann Russell, PhD, Principal Investigator — The Michener Institute for Education at UHN
Locations (1):
- Michener Chiropody Clinic, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No